CLINICAL TRIAL: NCT06381622
Title: The Effect of Combining Lidocaine and Ropivacaine on the Duration and Onset Time of an Ultrasound-guided Infraclavicular Brachial Plexus Nerve Block. a Randomized Controlled Trial
Brief Title: Combining Lidocaine and Ropivacaine for an Infraclavicular Brachial Plexus Nerve Block
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTA no: 2023-510028-63-00
Record Dates: First submitted 2024-04-12; First posted 2024-04-24 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-04

CONDITIONS: Nerve Block; Anesthesia, Local; Forearm Fracture; Surgery; Brachial Plexus Block
Keywords: Anesthetics, Local; Lidocaine; Ropivacaine
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group: Ropi-5 (Active Comparator): 30 ml Ropivacaine 5 mg/ml (equivalent to 150 mg Ropivacaine)
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution
- Intervention group 1: Ropi-5+Lido-20 (Experimental): 20 mL Ropivacaine 5 mg/ml + 10 mL Lidocaine-Epinephrine (20 mg + 5 µg) /ml (= 100 mg Ropivacaine + 200 mg Lidocaine)
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution; Drug: Lidocaine epinephrine
- Intervention group 2: Ropi-7.5+Lido-20 (Experimental): 20 mL Ropivacaine 7,5 mg/mL + 10 mL Lidocaine-Epinephrine (20 mg + 5 µg) /ml (= 150 mg Ropivacaine + 200 mg Lidocaine)
  Interventions: Drug: Lidocaine epinephrine; Drug: Ropivacaine 0.75% Injectable Solution

INTERVENTIONS:
Drug: Ropivacaine 0.5% Injectable Solution — 30 mL Ropivacaine 5 mg/mL (= 150 mg Ropivacaine)
  Arms: Control group: Ropi-5; Intervention group 1: Ropi-5+Lido-20
Drug: Lidocaine epinephrine — 20 mL Ropivacaine 5 mg/mL + 10 mL Lidocaine-Epinephrine (20 mg + 5 μg) / ml (= 100 mg Ropivacaine + 200 mg Lidocaine)
  Arms: Intervention group 1: Ropi-5+Lido-20; Intervention group 2: Ropi-7.5+Lido-20
Drug: Ropivacaine 0.75% Injectable Solution — 20 mL Ropivacaine 7,5 mg/mL + 10 mL Lidocaine-Epinephrine (20 mg + 5 μg)/mL (= 150 mg Ropivacaine + 200 mg Lidocaine)
  Arms: Intervention group 2: Ropi-7.5+Lido-20

SUMMARY:
The aim of the study is to investigate how the combination of ropivacaine (a slow onset, long duration local anesthetic) with lidocaine (a rapid onset, shorter duration local anesthetic) affects the onset and duration of a lateral infraclavicular plexus brachialis (LIC) block in patients undergoing non-acute hand surgery.

ELIGIBILITY:
Patient who have given written informed consent to participate in the study, after having understood it

Inclusion Criteria:

* Scheduled for non-acute hand surgery in regional anesthesia
* Scheduled for surgery on one of the following: 1) Antebrachium fractures or 2) Arthroplasty of a thumb base joint or 3) alloplasty of a thumb base joint

Exclusion Criteria:

* BMI > 40 kg/m2
* Weight < 60 kg
* Age < 18 years
* ASA physical status classification system grade > 3
* Allergy to experimental drugs
* Patients who cannot cooperate with the examinations or treatment
* Patients who do not understand or speak Danish
* Patients with peripheral or central neurological disease or nerve damage with neurological effect on the upper extremity, where surgery is required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-11-23 (Actual)

PRIMARY OUTCOMES:
Total time to breakthrough pain | 24 hours
  From the completion of the LIC block to first sensation of pain from the surgical area.

SECONDARY OUTCOMES:
The onset of sensory block | Until max 45 minutes
  From the completion of the LIC block to complete sensory blockade
  * Tested with refrigerator-cold glass vials.
  * A 3-point scale is used for cold sensation assessment: 1 point = normal sensation of cold, 2 points = reduced sensation of cold and 3 points = no cold sensation.
  * A complete sensory blockade is defined as all four tested nerves obtaining three points on the 3-point scale (no cold sensation).
  This outcome is measured until the complete block is obtained, but no longer than 45 minutes.
  - If a complete sensory block is not obtained after 45 minutes, the LIC block is viewed as a failed block.
Total duration of sensory blockade | 24 hours
  From the completion of the LIC block until the ending of sensory blockade
Total duration of motor blockade | 24 hours
  From the completion of the LIC block until the ending of motor blockade
Degree of motor blockade | At complete sensory blockade and otherwise 45 minutes after block performance
  Measured according to Manual Muscle Testing scale (4 point scale)
  * At the time of complete sensory blockade (defined as all four tested nerves obtaining three points on the 3-point scale (no cold sensation)), or if complete sensory blockade is not obtained, the degree of motor blockade is tested at 45 minutes.
  * Assessment is done using a 4-point Manual Muscle Testing Scale: 3 points = no difference, movement against resistance is possible, 2 points = a slight difference, movement against slight resistance is possible, 1 point = significant difference, movement is significantly compromised, 0 point = paralysis.

OTHER OUTCOMES:
Pain intensity at pain breakthrough | At pain breakthrough until a maximum of 24 hours after performed block.
  Via Numeric Rating Scale (NRS) 0 - 10 (0 = no pain; 10 = worst pain imaginable)
Duration of maximum pain intensity after the blockade has ended | After the blockade has ended until a maximum of 24 hours after performed block.
  Duration in hours:minutes
Occurence of adverse events (AE) and serious adverse events (SAE) | Follow up after 24 hours and 30 days
  Based on phone interviews and medical records
Failed blockade | Evaluated 30 minutes after completed surgery
  A block is viewed upon as failed if complete sensory block has not been achieved within 45 minutes or if supplemental local anaesthetic is needed before or during surgery.
The patient's experience of the treatment (patient satisfaction) | 24 hours
  Via Numeric Rating Scale (NRS) 0 - 10 (0 = very dissatisfied; 10 = very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Rothe, PhD, Principal Investigator — Nordsjællands Hospital, Københavns Universitet, Hillerød
Locations (1):
- Nordsjælland Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yousef S, Steensbaek MT, Bahuet AR, Knudsen RL, Harwood CD, Rosenstock CV, Andersen MF, Rothe C, Lange KHW, Norskov AK, Lundstrom LH. The effect of combining lidocaine and ropivacaine on the duration and onset time of an ultrasound-guided infraclavicular brachial plexus nerve block: A randomised controlled trial. Eur J Anaesthesiol. 2025 Dec 1;42(12):1046-1055. doi: 10.1097/EJA.0000000000002261. Epub 2025 Sep 1. PMID 40859881